CLINICAL TRIAL: NCT02117284
Title: Rubidium Elution System Performance Testing
Acronym: REST-PET
Status: Completed | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Jubilant DraxImage Inc. (Industry)
Responsible Party: Principal Investigator, Rob Beanlands, Chief, Division of Cardiology, Ottawa Heart Institute Research Corporation
Other Study IDs: 20130344
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: positron emission tomography (PET); Rubidium-82; myocardial perfusion imaging; automated elution system; controlled radioactivity delivery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary artery disease: All patients present to participating nuclear imaging facilities for diagnosis of CAD and/or risk stratification with Rubidium PET. Subjects will be enrolled according to the clinical indications listed in the approved Ruby-Fill product monograph.

SUMMARY:
Rubidium is a newly approved nuclear medicine imaging drug or 'tracer' used to look at blood flow in the heart. This tracer is given using a special pump called an 'elution system' which is considered investigational. This means the device is not yet approved by Health Canada for general use, but it has been approved for use in this study. It has been used routinely in this hospital since 2010.

The purpose of this study is to confirm proper operation of the pump. It may also help identify areas for future improvement. The study data may be used for safety reporting to the Ministry of Health or to Health Canada. The study will enroll 2,400 patients in 6 hospitals across Canada. The University of Ottawa Heart Institute (UOHI) will enroll up to 1,200 patients.

DETAILED DESCRIPTION:
Primary Objectives: To evaluate performance of the rubidium elution systems (RBES) manufactured by Jubilant DraxImage (JDI); specifically using the constant-activity-rate intravenous infusion of rubidium-82 from the Ruby-Fill™ generator for diagnostic imaging of myocardial perfusion with PET. The V3 elution system is more highly automated, therefore requiring fewer manual performance checks.

Hypotheses:

1. Performance: system operation using constant-activity infusion is adequate to achieve:

   1. elution activity (82Rb) bias < 5% (V2 and V3)
   2. elution activity (82Rb) imprecision < 5% (V2 and V3)
   3. elution time interval (30 s) bias < 5% (V2 only)
   4. elution success-rate reliability > 98% (failure-rate < 2%) (V2 and V3)
2. Daily Quality Assurance: testing procedures are adequate to document:

   1. Automated generator yield (82Rb) imprecision < 10% (V2 only)
   2. Automated generator breakthrough (82Sr, 85Sr) imprecision < 10% (V2 and V3)
   3. Manual generator yield (82Rb) imprecision < 10% (V2 only)
   4. Manual generator breakthrough (82Sr, 85Sr) imprecision < 10% (V2 only)
3. Monthly Quality Assurance: testing procedures are adequate to document:

   1. Dose calibrator non-linearity < 1% (V2 and V3)
   2. Dose calibrator constancy > 99% (instability < 1%) (V2 only)
   3. Dose calibrator bias < 10% (V2 only)
   4. Peristaltic pump calibration bias < 10% (V2 only) 2.2 Secondary Objectives: To evaluate the user documentation and training reliability for:
4. Installation of the Ruby-Fill generator and Ruby-Set tubing (V2 and V3)
5. Trouble-shooting and repair of system errors (e.g. high-pressure) (V2 and V3) 2.3 Tertiary Objective: To evaluate patient demographics or health status effects on system performance

ELIGIBILITY:
Inclusion Criteria:

All patients presenting to participating nuclear imaging facilities with Rb-82 PET for diagnosis and/or risk stratification for CAD (as listed in the approved Ruby-Fill product monograph), who are at least 18 years of age and have given informed consent or those who have consented to and are currently participating in an Ottawa Health Science Network Research Ethics Board (OHSN-REB) approved protocol utilizing Rb-82 PET will be eligible.

Exclusion Criteria:

* Patients with contraindications to stress radionuclide imaging including:
* Severe reactive airway disease;
* <3 days post myocardial infarction (MI) or acute coronary syndrome (ACS) presentation;
* Unstable crescendo angina;
* High grade atrioventricular (AV) block;
* Severe claustrophobia;
* Patients who are or may be pregnant will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients present to participating nuclear imaging facilities for diagnosis of CAD and/or risk stratification with Rubidium PET. Subjects will be enrolled according to the clinical indications listed in the approved Ruby-Fill product monograph.
Sampling Method: Probability Sample
Enrollment: 15800 (Actual)
Dates: Start 2014-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
System Performance: | 1 year
  System operation using constant-activity infusion is adequate to achieve:
  1. elution activity (82Rb) bias < 5% (V2 and V3)
  2. elution activity (82Rb) imprecision < 5% (V2 and V3)
  3. elution time interval (30 s) bias < 5% (V2 only)
  4. elution success-rate reliability > 98% (failure-rate < 2%) (V2 and V3)
Daily Quality Assurance: | 1 year
  System testing procedures are adequate to document:
  1. Automated generator yield (82Rb) imprecision < 10% (V2 only)
  2. Automated generator breakthrough (82Sr, 85Sr) imprecision < 10% (V2 and V3)
  3. Manual generator yield (82Rb) imprecision < 10% (V2 only)
  4. Manual generator breakthrough (82Sr, 85Sr) imprecision < 10% (V2 only)
Monthly Quality Assurance | 1 year
  System testing procedures are adequate to document:
  1. Dose calibrator non-linearity < 1% (V2 and V3)
  2. Dose calibrator constancy > 99% (instability < 1%) (V2 only)
  3. Dose calibrator bias < 10% (V2 only)
  4. Peristaltic pump calibration bias < 10% (V2 only)

SECONDARY OUTCOMES:
User documentation | 1 year
  To evaluate the user documentation and training reliability for:
  * Installation of the Ruby-Fill generator and Ruby-Set tubing (V2 and V3)
  * Trouble-shooting and repair of system errors (e.g. high-pressure) (V2 and V3)

CONTACTS AND LOCATIONS:
Overall Officials: Rob S Beanlands, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (4):
- Canada (4):
  - Hamilton Healath Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Background] Klein R, Adler A, Beanlands RS, Dekemp RA. Precision-controlled elution of a 82Sr/82Rb generator for cardiac perfusion imaging with positron emission tomography. Phys Med Biol. 2007 Feb 7;52(3):659-73. doi: 10.1088/0031-9155/52/3/009. Epub 2007 Jan 11. PMID 17228112